CLINICAL TRIAL: NCT02397434
Title: Adjuvant Radiotherapy After Cystectomy for Patients With Muscle Invasive Bladder Cancer: a Phase II Trial.
Brief Title: Adjuvant Radiotherapy After Cystectomy for Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/0630
Record Dates: First submitted 2014-11-19; First posted 2015-03-25 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Toxicity
Keywords: assessment of QOL (EORTC QLQ-C30)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adjuvant EBRT (Experimental): Radiation up to a median dose of 50 Gy in 25 fractions will be delivered with IMAT to the pelvic lymph node regions. If there is a positive surgical margin, the operative bladder bed will be included in the radiation field. A simultaneous integrated boost to positive lymph nodes will be delivered.
  Interventions: Radiation: Adjuvant EBRT

INTERVENTIONS:
Radiation: Adjuvant EBRT — Radiation up to a median dose of 50 Gy in 25 fractions will be delivered with IMAT to the pelvic lymph node regions. If there is a positive surgical margin, the operative bladder bed will be included in the radiation field. A simultaneous integrated boost to positive lymph nodes will be delivered.

SUMMARY:
A radical cystectomy + extended pelvic lymph node dissection is considered to be the treatment of choice for patients with muscle invasive bladder cancer (MIBC). Despite this aggressive treatment the outcome is poor and ultimately, 30% of the patients with ≥pT3 tumors develop a pelvic recurrence. One- and 2-years survival for patients developing a local recurrence after cystectomy is only 8% and 3% respectively, with a median survival of <4 months. For patients with lymph node recurrence prognosis is somewhat better, but nevertheless still disappointing with reported 1- and 2 years survival of 42% and 11% respectively. The investigators hypothesize that an earlier implementation of external beam radiotherapy (EBRT) i.e. in the adjuvant setting, will prevent local and lymph node recurrence and improve disease free- and overall survival as local recurrence is linked to the development of distant metastasis. Adjuvant EBRT was tested in a prospective randomized trial and resulted in a 20% increase in 5-year disease free survival. Despite those impressive results, severe intestinal toxicity rates hampered the enthusiasm to use adjuvant EBRT, till now. In the last decade, great technological advancements in EBRT planning, such as intensity modulated arc therapy (IMAT), and positioning have been realised. This has resulted in a better coverage of the target volume while sparing normal tissue (mainly small bowel) and in a more precise delivery of the EBRT. Therefore, it is desirable to reconsider the use of adjuvant EBRT in selected MIBC patients.

DETAILED DESCRIPTION:
The investigators plan to perform a prospective phase 2 study including 76 patients.

Radiation up to a median dose of 50 Gy in 25 fractions will be delivered with IMAT to the pelvic lymph node regions. If there is a positive surgical margin, the operative bladder bed will be included in the radiation field. A simultaneous integrated boost to 64 Gy to the positive lymph nodes will be delivered. Pathological evaluation on cystectomy specimen includes: tumor stage and grade, area of necrosis (absolute and relative), micro vessel density, epidermal growth factor receptor.

ELIGIBILITY:
Inclusion Criteria: muscle invasive bladder cancer with:

* ≥ pathological tumor stage (p)T3 stage + presence of lymphovascular invasion on pathological examination
* pT4
* <10 lymph nodes removed
* positive lymph nodes
* positive surgical margins

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in acute Radiation Therapy Oncology Group (RTOG) toxicity | last day of radiotherapy, 1 month and 3 months after last day of EBRT

SECONDARY OUTCOMES:
change from baseline in late RTOG toxicity | at 6,9, 12, 18 and 24months after last day of EBRT
change from baseline in local control | at 6,9, 12, 18 and 24months after last day of EBRT
disease free survival | at 6,9, 12, 18 and 24months after last day of EBRT
overall survival | at 6,9, 12, 18 and 24months after last day of EBRT

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Fonteyne, Principal Investigator — University Hospital, Ghent
Locations (1):
- Dept of Radiotherapy, University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Fonteyne V, Dirix P, Junius S, Rammant E, Ost P, De Meerleer G, Swimberghe M, Decaestecker K. Adjuvant radiotherapy after radical cystectomy for patients with muscle invasive bladder cancer: a phase II trial. BMC Cancer. 2017 May 2;17(1):308. doi: 10.1186/s12885-017-3302-9. PMID 28464906